CLINICAL TRIAL: NCT03773263
Title: New Application of Oocyte Sequential Culture and in Vitro Muturation System for Infertility Patients With Polycystic Ovary Syndrome: a Multi-center Prospective Randomized Clinical Trial
Brief Title: New Application of Sequential in Vitro Muturation System for Infertility Patients With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Hospital for Reproductive Medicine Affiliated to Shandong University (Unknown); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Yanhong Deng, doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: newivf20181206
Record Dates: First submitted 2018-12-08; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: sequential IVM system; PCOS; infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sequential oocyte IVM group (Experimental): From day 7~9 of the menstrual cycle, 225 IU HMG (Menotrophins for Injection) per day will be administrated for 3 days. COCs were removed from aspirated follicular fluid and transferred into HEPES-buffered collection medium. The immature oocytes will be cultured in sequential IVM medium 1 for 6 hours (37℃, 5% CO2), and removed into sequential IVM medium 2 for further cultivation. After 24 and 40 hours cultivation, the mature oocytes will be fertilized by intracytoplasmic sperm injection (ICSI). Two of the D3 embryos (if available) which graded as top-quality embryo will be vitrified and the rest of embryos will be cultivated extendedly. Thawed embryo transfer (TET) will give preference to D3 embryos and carried out with a hormone replacement cycle.
  Interventions: Drug: sequential IVM system; Procedure: intracytoplasmic sperm injection (ICSI); Procedure: Thawed embryo transfer (TET)
- traditional oocyte IVM group (Active Comparator): From day 7~9 of the menstrual cycle, 225 IU HMG (Menotrophins for Injection) per day will be administrated for 3 days. On the day of ovulation, COCs were aspirated and the immature oocytes will be cultured in traditional standard oocyte IVM system (Sage). 30 and 44 hours after cultivation, the maturity of oocytes will be assessed and the mature oocytes will be fertilized by intracytoplasmic sperm injection (ICSI). Two of the D3 embryos (if available) which graded as top-quality embryo will be vitrified and the rest of embryos will be cultivated extendedly. Thawed embryo transfer (TET) will give preference to D3 embryos and carried out with a hormone replacement cycle. If biochemical pregnancy is not achieved, thawed blastocysts transfer will be performed.
  Interventions: Procedure: intracytoplasmic sperm injection (ICSI); Procedure: Thawed embryo transfer (TET); Drug: traditional IVM system

INTERVENTIONS:
Drug: sequential IVM system — The immature oocytes will be cultured in sequential oocyte IVM medium 1 for 6 hours (37℃, 5% CO2). After flushed 3 times, COCs were removed into sequential oocyte IVM medium 2 for further cultivation.
  Arms: sequential oocyte IVM group
Procedure: intracytoplasmic sperm injection (ICSI) — intracytoplasmic sperm injection (ICSI)
Procedure: Thawed embryo transfer (TET) — Patients administrates oestrogen (Progynova) 3mg twice a day for 10 to 12 days. From the day when endometrium reach a thickness of 8 mm and above, luteal phase support will be given with 10 mg progesterone (Dydrogesterone Tablets,) triple per day and utrogestan (Laboratories Besins International, Paris, France) 0.2g triple per day, until 14 days after embryo transfer.
Drug: traditional IVM system — COCs were aspirated and the immature oocytes will be cultured in traditional standard oocyte IVM system (Sage). 30 and 44 hours after cultivation, the maturity of oocytes will be assessed.
  Other Names: sage
  Arms: traditional oocyte IVM group

SUMMARY:
Oocyte in vitro maturation (IVM) is an artificial reproductive technologies (ART) in which cumulus-oocyte complex (COC) are collected at the immature germinal vesicle (GV) stage from unstimulated or FSH-primed ovaries and matured in vitro before fertilization. IVM has been proposed as a more patient-friendly ART alternative to conventional IVF. Contrary to IVF, IVM is the only ART method with no cases of OHSS reported. Hence, patients with PCOS represent the major target population for IVM treatment.

In clinical practice of standard IVM, COCs are aspirated from unstimulated or mildly stimulated ovaries and rapidly removed from the meiotic-inhibiting influence of the follicle and the follicular fluid. Regardless of in vitro gonadotrophin treatment, oocytes mature spontaneously in vitro, hence undergoing meiotic resumption in the absence of the usual elaborate cascade of endocrine and paracrine molecular signals that induce maturation in vivo. As such, the maturation of oocytes by standard IVM techniques is an artefact that compromises subsequent oocyte developmental competence. Numbers of studies have been proposed to improve the efficiency of IVM system. Synchronization of meiotic and cytoplasmic maturation in antral oocytes arrested at the immature GV-stage remains a major challenge and is of fundamental importance for successful fertilization. High intra-oocyte levels of cyclic adenosine monophosphate (cAMP), is crucial to maintain the nearly fully-grown oocytes under meiotic arrest and to induce oocyte maturation. Research in animal models has indicated that a non-physiological drop of cAMP levels in the oocyte results in asynchronous nuclear and cytoplasmic maturation.

Investigators have reported the development of a novel in vitro simulated sequential oocyte maturation system. Critical to success of the approach is a pre-IVM phase that generates a rapid increase in COC cAMP levels. Secondly, the system utilizes an extended IVM phase containing sufficient FSH to drive meiotic induction in the presence of a type-3 PDE inhibitor. The high levels of cAMP in the oocyte and the induced nature of oocyte maturation mimics some of the key, newly characterized molecular signals that occur during oocyte maturation in vivo. Technical and conceptual elements were first developed using mouse, bovine and human COCs. Investigators propose a randomized clinical trial to compare a novel sequential culture system with the traditional standard oocyte IVM system for PCOS patients.

DETAILED DESCRIPTION:
A multi-center, prospective, randomized clinical trial will be conducted, of comparing sequential oocyte IVM system with traditional oocyte IVM system for high OHSS risk PCOS patients (AMH>5.6ng/ml). The inclusion criteria will be infertile patients diagnosed by the Chinese PCOS criteria, aged below 35 years, and without other known factors interfere reproductive or metabolic functions. 300 PCOS patients will be included and randomized into either of two groups: group A will administrate sequential oocyte IVM system and group B will administrate traditional standard oocyte IVM system. The comparison will be made between groups, and both groups are conducted with the HMG administration and embryo vitrification freezing. The primary outcome of the study is live birth rate. The embryo development and pregnancy outcomes will be followed up and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Women age ≤35 years;
2. AMH level ≥5.6ng/ml;
3. Women diagnosed as PCOS according to Chinese PCOS diagnosis criteria;
4. Written informed consent.

Exclusion Criteria:

* Women who diagnosed as uterus abnormality, adenomyosis, submucous myoma, intrauterine adhesion;
* Women who diagnosed as untreated hydrosalpinx;
* Women who had underwent unilateral ovariectomy;
* Women with medical condition that represent contraindication to assisted reproductive technology or pregnancy;
* Women or their partner with abnormal chromosome karyotype;
* Male partner with oligoasthenozoospermia or obstructive azoospermia;
* Male partner whose sperm is collected by surgery;
* Subjects are found breach the inclusion criteria, or in accordance with exclusion criteria during the test, excluded;
* Patients request withdrawal and exit the trial because adverse events occur during the trial.

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7 weeks gestation
  The fetal heart beat in an intrauterine gestational sac under ultrasound will be defined as clinical pregnancy.

SECONDARY OUTCOMES:
Oocyte maturation rate | 30 and 46 hours after oocyte retrieval
  Oocyte maturation rate (%): number of MII oocytes/ number of oocytes retrieved.
Fertilization rate | 30 and 46 hours after oocyte retrieval
  Fertilization rate (%): number of oocytes fertilized/ number of oocytes retrieved.
Cleavage rate | 24 hours after ICSI
  Cleavage rate (%): number of cleavages/ number of 2PN embryos.
Day 3 embryo rate | 72 hours after ICSI
  Day 3 embryo rate (%): number of Day 3 embryos / number of 2PN embryos.
Good quality embryo rate at cleavage-stage | 72 hours after ICSI
  Good quality embryo rate at cleavage-stage (%): number of good quality embryos at cleavage-stage / number of 2PN embryos.
Number of cycles with available embryo | 72 hours after ICSI
  Available embryos will be defined as three days after oocyte retrieval with containing more than 4 cells and grade 1 to 2 or containing 4 cells with a grade of 1.
Blastulation rate | 144 hours after ICSI
  Blastulation rate (%): number of blastocysts / number of 2PN embryos.
Biochemical pregnancy rate | 4 weeks gestation
  A serum β-hCG level above 5 IU/L, which is performed 12 days after embryos transfer, will be defined as biochemical pregnancy.
Implantation rate | 7 weeks gestation
  The implantation rate will be defined as the number of gestational sacs seen on the ultrasound divided by the total number of embryos transferred.
Miscarriage rate (at first trimester) | 28 weeks gestation in maximum
  Miscarriage at first trimester will be defined by any positive pregnancy test that result in a loss of pregnancy before 12 weeks gestation.
Cumulative pregnancy rate | 1-2year
  Cumulative pregnancy rate will be defined as clinical pregnancies with intrauterine fetal heart beat detected divided by the number of retrieval cycles whose embryos are all transferred.
Preterm birth rate | 1-2year
  Preterm birth means the baby is born before the 37th week of pregnancy in China.
Newborn birth weight | 1-2year
  Newborn birth weight
Neonatal complication rate | within one month after labor
  We will collect complications that occur in the neonate including admission to the neonatal intensive care unit (NICU), hospitalization, etc.
Live birth rate | 1-2year
  Live birth rate(%): number of live birth/ transferred cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-yan Liang, M.D. & Ph.D, Study Director — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (5):
- China (5):
  - The Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Reproductive medical hospital affiliated to Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Tenth People's Hospital of Tongji University, Shanghai